CLINICAL TRIAL: NCT02415348
Title: The Use of Fibroscan to Assess Liver Fibrosis in Patients With Cardiac Pacemakers and/or Implantable Cardioverter-Defibrillators
Brief Title: The Use of Fibroscan to Assess Liver Fibrosis in Patients With Cardiac Pacemakers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Bio 15-35
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan (Experimental): Fibroscan under simultaneous cardiac monitoring
  Interventions: Device: Fibroscan

INTERVENTIONS:
Device: Fibroscan

SUMMARY:
This study is designed to determine if the Fibroscan (Echosens, Paris), a non-invasive, ultrasound-based device used to estimate fibrosis in patients with chronic liver disease, interferes with implanted cardiac pacemaker and/or implantable cardioverter-defibrillators. Recruitment consists of a total of 200 outpatients undergoing routine pacemaker interrogation at a teaching-hospital pacemaker clinic.

DETAILED DESCRIPTION:
Assessment of liver fibrosis in patients with chronic liver diseases provides staging and prognostic information critical in establishing treatment priorities. The gold standard evaluation of liver fibrosis is hampered by the invasive nature of liver biopsies. FibroScan is a non-invasive alternative that has been extensively validated in chronic hepatitis C, chronic hepatitis B, alcoholic liver disease, and non- alcoholic fatty liver disease patients.

To avoid unknown risks of potential interaction, the manufacturer have advised against the use of the device in patients with active implantable medical device including cardiac pacemaker and/or implantable cardioverter-defibrillators(ICD). Review of the literature showed that these two population have been specifically excluded in all previously reported studies.

At the time of writing, no specific reports have demonstrated either safety or potential harm of the FibroScan in patients with pacemaker/ICD. Given the proven benefit of the FibroScan in chronic liver disease and the current policy of excluding patients with pacemaker/ICD in clinical practice, this study aims to formally evaluate the safe use of the FibroScan in this population within the controlled environment of a pacemaker lab.

ELIGIBILITY:
Inclusion Criteria:

-Any outpatient undergoing routine pacemaker interrogation at pacemaker clinic

Exclusion Criteria:

* Pregnancy
* BMI>35
* Person with active implantable medical devices other than cardiac pacemaker and/or ICD
* Person who are unable to tolerate lying flat for the FibroScan examination.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Pacemaker/ICD malfunction | 30 min
Type of Pacemaker/ICD malfunction | 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Worobetz, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada